CLINICAL TRIAL: NCT01452841
Title: Efficiency of Daily Grapefruit Exposure in Reducing Body Weight and Inflammatory Markers
Brief Title: A Grapefruit Feeding Trial in Healthy, Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09-0695-02
Record Dates: First submitted 2011-07-21; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Weight Loss; Obesity; Cardiovascular Risk Factors
Keywords: grapefruit; weight loss; blood pressure; lipids; inflammation
MeSH Terms: conditions — Weight Loss; Obesity; Inflammation | interventions — grapefruit seed extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grapefruit Consumption (Experimental)
  Interventions: Other: Grapefruit
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Grapefruit — 1.5 Rio Red Grapefruit consumed daily for 6 weeks
  Arms: Grapefruit Consumption
Other: Control — Participants followed a diet low in bioactive rich fruits and vegetables and avoided citrus for six weeks
  Arms: Control

SUMMARY:
Folklore has suggested that consuming grapefruit may promote weight control. Sparse data exist to support this hypothesis, though there is some evidence of health promotional effects regarding blood pressure and lipid profiles. The aims of this randomized controlled trial are to determine the role of grapefruit in:

1. Reducing weight
2. Reducing blood pressure
3. Reducing inflammation
4. Improving the lipid profile.

The investigators hypothesize that six weeks of daily consumption of grapefruit will reduce weight, blood pressure, and inflammation while improving the lipid profile in overweight, healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults, men and premenopausal women
* BMI: 25-45 kg/m2
* Willing to maintain current exercise regimen (not to exceed 10 hours/week)
* Willing to follow a diet low in bioactive rich fruits and vegetables and with no citrus

Exclusion Criteria:

* History of chronic disease
* Metabolic disease
* Inflammatory disease
* High cholesterol (>225 mg/dL)
* Smoker
* Taking medications metabolized by the Cytochrome P450 3A enzyme
* History of alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Weight reduction | 6 weeks
  Participants consumed 1/2 grapefruit before each meal (1.5 grapefruit per day) for six weeks. Weight was measured before and after grapefruit consumption to assess weight change. Weight change was considered statistically significant at p<0.05.

SECONDARY OUTCOMES:
Blood pressure reduction | 6 weeks
  Previous studies in animals and humans consuming citrus have resulted in reductions in blood pressure, though no direct effect of grapefruit has ever been demonstrated. Blood pressure was measured at baseline and after the 6 week intervention period (consuming either the control diet or supplementing the diet with 1/2 grapefruit before each meal).
Lipid Profile Improvements | 6 weeks
  Previous studies in humans and animal models consuming grapefruit or grapefruit bioactives have shown reductions in triglycerides, LDL, and total cholesterol and increases in circulating HDL. These parameters were measured via a common point-of-care system, LDX Cholestech. Lipids were measured at baseline and after the 6 week intervention period (consuming either the control diet or supplementing the diet with 1/2 grapefruit before each meal).
Reductions in markers of chronic inflammation | 6 weeks
  Markers of chronic inflammation, which are also associated with endothelial dysfunction and heart disease, like tumor necrosis factor alpha (TNFalpha), interleukin-1beta (IL-1beta), and soluble vascular cellular adhesion molecule-1 (sV-CAM1) were measured. Inflammatory markers were measured at baseline and after the 6 week intervention period (consuming either the control diet or supplementing the diet with 1/2 grapefruit before each meal).

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Thomson, PhD, RD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States